CLINICAL TRIAL: NCT01586910
Title: Surgical Replacement and Transcatheter Aortic Valve Implantation (SURTAVI)
Brief Title: Safety and Efficacy Study of the Medtronic CoreValve® System in the Treatment of Severe, Symptomatic Aortic Stenosis in Intermediate Risk Subjects Who Need Aortic Valve Replacement (SURTAVI).
Acronym: SURTAVI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDE #G120169
Record Dates: First submitted 2012-04-24; First posted 2012-04-27 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Medtronic CoreValve® System TAVI (Experimental): Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Device: Medtronic CoreValve® Evolut R System Transcatheter Aortic Valve Implantation (TAVI)
- SAVR (Active Comparator): Surgical Aortic Valve Replacement (SAVR)
  Interventions: Procedure: Surgical Aortic Valve Replacement (SAVR)

INTERVENTIONS:
Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Arms: Medtronic CoreValve® System TAVI
Procedure: Surgical Aortic Valve Replacement (SAVR)
  Arms: SAVR
Device: Medtronic CoreValve® Evolut R System Transcatheter Aortic Valve Implantation (TAVI)
  Arms: Medtronic CoreValve® System TAVI

SUMMARY:
The purpose of the study is to investigate the safety and efficacy of transcatheter aortic valve implantation (TAVI) in patients with severe, symptomatic Aortic Stenosis (AS) at intermediate surgical risk by randomizing patients to either Surgical Aortic Valve Replacement (SAVR) or TAVI with the Medtronic CoreValve® System.

Single Arm: The purpose of this trial is to evaluate the safety and effectiveness of transcatheter aortic valve implementation (TAVI) in patients with severe symptomatic Aortic Stenosis (AS) at intermediate surgical risk with TAVI. This is a non-randomized phase of the pivotal clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have co-morbidities such that Heart Team agrees predicted risk of operative mortality is ≥3% and <15% at 30 days (Intermediate Clinical Risk classification). Heart team evaluation of clinical surgical mortality risk for each patient includes the calculated STS score for predicted risk of surgical mortality augmented by consideration of the overall clinical status and co-morbidities unmeasured by the STS risk calculation;
* Heart Team unanimously agree on treatment proposal and eligibility for randomization* based on their clinical judgement (including anatomy assessment, risk factors, etc.);
* Subject has severe aortic stenosis presenting with;

  1. Critical aortic valve area defined as an initial aortic valve area of ≤1.0cm2 or aortic valve area index < 0.6cm2/m2 AND
  2. Mean gradient > 40mmHg or Vmax > 4m/sec by resting echocardiogram or simultaneous pressure recordings at cardiac catherization [or with dobutamine stress, if subject has left ventricular ejection fraction (LVEF) <55%] or velocity ratio < 0.25;
* Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater;
* Subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits;
* Subject meets the legal minimum age to provide informed consent based on local regulatory requirements;

Exclusion Criteria:

* Subject has refused surgical aortic valve replacement (SAVR) as a treatment option; (not applicable for Single Arm)
* Any condition considered a contraindication for placement of a bioprosthetic valve (i.e., subject requires a mechanical valve);
* A known hypersensitivity or contraindication to all anticoagulation/antiplatelet regimens (or inability to be anticoagulated for the index procedure), nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated;
* Blood dyscrasias as defined: leukopenia (WBC <1000mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy;
* Ongoing sepsis, including active endocarditis;
* Any condition considered a contraindication to extracorporeal assistance;
* Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to randomization* (Subjects with recent placement of drug eluting stent(s) should be assessed for ability to safely proceed with SAVR within the protocol timeframe);
* Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within six weeks of randomization*;
* Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support;
* Recent (within 6 months of randomization*) cerebrovascular accident (CVA) or transient ischemic attack (TIA);
* Active gastrointestinal (GI) bleeding that would preclude anticoagulation;
* Subject refuses a blood transfusion;
* Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits);
* Multivessel coronary artery disease with a Syntax score >22 and/or unprotected left main coronary artery (Syntax score calculation is not required for patients with history of previous revascularization if repeat revascularization is not planned);
* Estimated life expectancy of less than 24 months due to associated non-cardiac comorbid conditions;
* Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams;
* Currently participating in an investigational drug or another device trial (excluding registries);
* Evidence of an acute myocardial infarction ≤30 days before the index procedure;
* Need for emergency surgery for any reason;
* True porcelain aorta (i.e. Heart Team agrees the aorta is not clampable for SAVR);
* Extensive mediastinal radiation;
* Liver failure (Child-C);
* Reduced ventricular function with left ventricular ejection fraction (LVEF) <20% as measured by resting echocardiogram;
* Uncontrolled atrial fibrillation (e.g. resting heart rate > 120 bpm);
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up requirements;
* End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min;
* Pulmonary Hypertension (systolic pressure> 80mmHg);
* Severe Chronic Obstructive Pulmonary Disease (COPD) demonstrated by Forced Expiratory Volume (FEV1) < 750cc;
* Frailty assessments identify:

  1. Subject is < 80 years of age and three or more of the following apply
  2. Subject is ≥ 80 years of age and two or more of the following apply

     * Wheelchair bound
     * Resides in an institutional care facility (e.g., nursing home, skilled care center)
     * Body Mass Index < 20 kg/m2
     * Grip Strength < 16 kg
     * Katz Index Score ≤ 4
     * Albumin < 3.5 g/dL;
* Marfan syndrome or other known connective tissue disease that would necessitate aortic root replacement/intervention; (Not applicable for Single Arm)

Note: Additional anatomical and vascular exclusion criteria may apply.

Note: * For purposes of the single arm phase of the trial, "randomization" will refer to trial enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1746 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2026-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, MD, PhD, Principal Investigator — Bern University Hospital; Rüdiger Lange, MD, PhD, Principal Investigator — Deutsches Herzzentrum München; Thomas Walther, MD, PhD, Principal Investigator — Kerckhoff Klinik; Michael J. Reardon, MD, Principal Investigator — The Methodist Hospital Research Institute; David H. Adams, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Nicolas M. Van Mieghem, MD, Study Chair — Erasmus Medical Center; Patrick W. Serruys, MD, PhD, Study Chair — National Heart & Lung Institute of Imperial College in London
Locations (86):
- United States (65):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Hollywood, California
  - Scripps Green Hospital, La Jolla, California
  - Keck Medical Center of USC, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Southern California Permenente Medical Group, Pasadena, California
  - Stanford University Medical Center, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Miami, Coral Gables, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare, Inc., Atlanta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Loyola University of Chicago, Maywood, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center / Mercy Medical Center, West Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Cardiovascular Institute of the South, Houma, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Inc., Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Detroit Medical Center, Detroit, Michigan
  - Henry Ford, Detroit, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Abbott NW - MN Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic - St. Mary's Hospital, Rochester, Minnesota
  - Saint Luke's Hospital/MAHI, Kansas City, Missouri
  - Alegent Creighton Health Research Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - New York University School of Medicine, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The OhioHealth Research Institute, Columbus, Ohio
  - Oklahoma Heart Institute, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Wormleysburg, Pennsylvania
  - Stern Cardiovascular, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - The Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - The Heart Hospital - Baylor Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Vermont, Burlington, Vermont
  - Sentara Cardiovascular, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (5):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Toronto General Hospital (University Health Network), Toronto, Ontario
  - McGill University Health Center - Royal Victoria Hospital, Montreal, Quebec
  - Montreal Heart Institute, Montreal
- Rigshospitalet, Copenhagen, Denmark
- Germany (3):
  - Universitäts-Herzzentrum Freiburg • Bad Krozingen, Bad Krozingen
  - Universitätsklinikum Bonn, Bonn
  - Deutsches Herzzentrum Muenchen, Munich
- Netherlands (4):
  - Amphia Hospital Breda, Breda
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Antonius Hospital, R & D Cardiology, Nieuwegein
  - Erasmus Medical Center - Rotterdam, Rotterdam
- Spain (2):
  - Servicio de Cardiologia del Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
- Karolinska Universitetssjukhuset Stockholm, Stockholm, Sweden
- Switzerland (2):
  - Bern University Hospital, Bern
  - Universitatsspital Zurich, Zurich
- United Kingdom (3):
  - Leeds General Infirmary, Leeds
  - Glenfield Hospital, Leicester, UK, Leicester
  - St. George's Hospital London, London

REFERENCES:
- [Derived] Klautz RJM, Rao V, Reardon MJ, Deeb GM, Dagenais F, Moront MG, Little SH, Labrousse L, Patel HJ, Ito S, Li S, Sabik JF 3rd, Oh JK. Examining the typical hemodynamic performance of nearly 3000 modern surgical aortic bioprostheses. Eur J Cardiothorac Surg. 2024 May 3;65(5):ezae122. doi: 10.1093/ejcts/ezae122. PMID 38710669
- [Derived] Kleiman NS, Van Mieghem NM, Reardon MJ, Gada H, Mumtaz M, Olsen PS, Heiser J, Merhi W, Chetcuti S, Deeb GM, Chawla A, Kiaii B, Teefy P, Chu MWA, Yakubov SJ, Windecker S, Althouse AD, Baron SJ. Quality of Life 5 Years Following Transfemoral TAVR or SAVR in Intermediate Risk Patients. JACC Cardiovasc Interv. 2024 Apr 22;17(8):979-988. doi: 10.1016/j.jcin.2024.02.014. PMID 38658126
- [Derived] O'Hair D, Yakubov SJ, Grubb KJ, Oh JK, Ito S, Deeb GM, Van Mieghem NM, Adams DH, Bajwa T, Kleiman NS, Chetcuti S, Sondergaard L, Gada H, Mumtaz M, Heiser J, Merhi WM, Petrossian G, Robinson N, Tang GHL, Rovin JD, Little SH, Jain R, Verdoliva S, Hanson T, Li S, Popma JJ, Reardon MJ. Structural Valve Deterioration After Self-Expanding Transcatheter or Surgical Aortic Valve Implantation in Patients at Intermediate or High Risk. JAMA Cardiol. 2023 Feb 1;8(2):111-119. doi: 10.1001/jamacardio.2022.4627. PMID 36515976
- [Derived] Tuttle MK, Kiaii B, Van Mieghem NM, Laham RJ, Deeb GM, Windecker S, Chetcuti S, Yakubov SJ, Chawla A, Hockmuth D, Teefy P, Li S, Reardon MJ. Functional Status After Transcatheter and Surgical Aortic Valve Replacement: 2-Year Analysis From the SURTAVI Trial. JACC Cardiovasc Interv. 2022 Apr 11;15(7):728-738. doi: 10.1016/j.jcin.2022.01.284. PMID 35393106
- [Derived] Lanz J, Reardon MJ, Pilgrim T, Stortecky S, Deeb GM, Chetcuti S, Yakubov SJ, Gleason TG, Huang J, Windecker S. Incidence and Outcomes of Infective Endocarditis After Transcatheter or Surgical Aortic Valve Replacement. J Am Heart Assoc. 2021 Oct 5;10(19):e020368. doi: 10.1161/JAHA.120.020368. Epub 2021 Sep 28. PMID 34581194
- [Derived] Mumtaz M, Wyler von Ballmoos MC, Deeb GM, Popma JJ, Van Mieghem NM, Kleiman NS, Gleason TG, Chawla A, Hockmuth D, Zorn GL 3rd, Tadros P, Li S, Reardon MJ. The Impact of Transfusions on Mortality After Transcatheter or Surgical Aortic Valve Replacement. Ann Thorac Surg. 2021 Sep;112(3):778-785. doi: 10.1016/j.athoracsur.2020.09.031. Epub 2020 Nov 17. PMID 33217396
- [Derived] Attizzani GF, Dallan LAP, Markowitz A, Yakubov SJ, Deeb GM, Reardon MJ, Forrest JK, Mangi AA, Huang J, Popma JJ. Impact of Repositioning on Outcomes Following Transcatheter Aortic Valve Replacement With a Self-Expandable Valve. JACC Cardiovasc Interv. 2020 Aug 10;13(15):1816-1824. doi: 10.1016/j.jcin.2020.04.028. PMID 32763073
- [Derived] Yakubov SJ, Van Mieghem NM, Reardon MJ, Serruys PW, Gada H, Mumtaz M, Deeb GM, Kodali S, George I, Windecker S, Kleiman N, Chetcuti SJ, Sanchez C, Dauerman HL, Li S, Popma JJ. Propensity-Matched Comparison of Evolut-R Transcatheter Aortic Valve Implantation With Surgery in Intermediate-Risk Patients (from the SURTAVI Trial). Am J Cardiol. 2020 Sep 15;131:82-90. doi: 10.1016/j.amjcard.2020.06.051. Epub 2020 Jun 29. PMID 32723555
- [Derived] Van Mieghem NM, Reardon MJ, Yakubov SJ, Heiser J, Merhi W, Windecker S, Makkar RR, Cheng W, Robbins M, Fail P, Feinberg E 2nd, Stoler RC, Hebeler R, Serruys PW, Popma JJ. Clinical outcomes of TAVI or SAVR in men and women with aortic stenosis at intermediate operative risk: a post hoc analysis of the randomised SURTAVI trial. EuroIntervention. 2020 Nov 20;16(10):833-841. doi: 10.4244/EIJ-D-20-00303. PMID 32715995
- [Derived] Lindman BR, Goel K, Bermejo J, Beckman J, O'Leary J, Barker CM, Kaiser C, Cavalcante JL, Elmariah S, Huang J, Hickey GL, Adams DH, Popma JJ, Reardon MJ. Lower Blood Pressure After Transcatheter or Surgical Aortic Valve Replacement is Associated with Increased Mortality. J Am Heart Assoc. 2019 Nov 5;8(21):e014020. doi: 10.1161/JAHA.119.014020. Epub 2019 Oct 31. PMID 31665959
- [Derived] Sondergaard L, Popma JJ, Reardon MJ, Van Mieghem NM, Deeb GM, Kodali S, George I, Williams MR, Yakubov SJ, Kappetein AP, Serruys PW, Grube E, Schiltgen MB, Chang Y, Engstrom T. Comparison of a Complete Percutaneous Versus Surgical Approach to Aortic Valve Replacement and Revascularization in Patients at Intermediate Surgical Risk: Results From the Randomized SURTAVI Trial. Circulation. 2019 Oct 15;140(16):1296-1305. doi: 10.1161/CIRCULATIONAHA.118.039564. Epub 2019 Sep 3. PMID 31476897
- [Derived] Reardon MJ, Heijmen RH, Van Mieghem NM, Williams MR, Yakubov SJ, Watson D, Kleiman NS, Conte J, Chawla A, Hockmuth D, Petrossian G, Robinson N, Kappetein AP, Li S, Popma JJ. Comparison of Outcomes After Transcatheter vs Surgical Aortic Valve Replacement Among Patients at Intermediate Operative Risk With a History of Coronary Artery Bypass Graft Surgery: A Post Hoc Analysis of the SURTAVI Randomized Clinical Trial. JAMA Cardiol. 2019 Aug 1;4(8):810-814. doi: 10.1001/jamacardio.2019.1856. PMID 31215985
- [Derived] Head SJ, Reardon MJ, Deeb GM, Van Mieghem NM, Popma JJ, Gleason TG, Williams MR, Radhakrishnan S, Fremes S, Oh JK, Chang Y, Boulware MJ, Kappetein AP. Computed Tomography-Based Indexed Aortic Annulus Size to Predict Prosthesis-Patient Mismatch. Circ Cardiovasc Interv. 2019 Apr;12(4):e007396. doi: 10.1161/CIRCINTERVENTIONS.118.007396. PMID 30929507
- [Derived] Durko AP, Reardon MJ, Kleiman NS, Popma JJ, Van Mieghem NM, Gleason TG, Bajwa T, O'Hair D, Brown DL, Ryan WH, Chang Y, De Leon SD, Kappetein AP. Neurological Complications After Transcatheter Versus Surgical Aortic Valve Replacement in Intermediate-Risk Patients. J Am Coll Cardiol. 2018 Oct 30;72(18):2109-2119. doi: 10.1016/j.jacc.2018.07.093. PMID 30360820
- [Derived] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Derived] Haussig S, Linke A. Patient selection for TAVI 2015 - TAVI in low-risk patients: fact or fiction? EuroIntervention. 2015 Sep;11 Suppl W:W86-91. doi: 10.4244/EIJV11SWA27. PMID 26384204
- [Derived] Piazza N, Kalesan B, van Mieghem N, Head S, Wenaweser P, Carrel TP, Bleiziffer S, de Jaegere PP, Gahl B, Anderson RH, Kappetein AP, Lange R, Serruys PW, Windecker S, Juni P. A 3-center comparison of 1-year mortality outcomes between transcatheter aortic valve implantation and surgical aortic valve replacement on the basis of propensity score matching among intermediate-risk surgical patients. JACC Cardiovasc Interv. 2013 May;6(5):443-51. doi: 10.1016/j.jcin.2013.01.136. PMID 23702009

RESULTS

PARTICIPANT FLOW:
Groups:
- Medtronic CoreValve® System TAVI: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® Evolut R System Transcatheter Aortic Valve Implantation (TAVI)
Period: Overall Study
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Started | 879 | 867
Completed | 864 | 796
Not Completed | 15 | 71
Not completed — Death | 4 | 4
Not completed — Withdrawal by Subject | 6 | 43
Not completed — Physician withdrew Subject | 5 | 24

BASELINE CHARACTERISTICS:
Population: mITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Medtronic CoreValve® System TAVI | SAVR | Total
Number analyzed (Participants) | 864 | 796 | 1660
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
  years | 79.9 (6.2) | 79.7 (6.1) | 79.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
  Participants
    Female | 366 | 358 | 724
    Male | 498 | 438 | 936
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data from three race categories (Asian, Black/African American/ Hispanic or Latino Ethnicity) were collected in the study.
  Participants
    number analyzed (Participants) | 43 | 50 | 93
    Asian | 7 | 6 | 13
    Black/African American | 18 | 21 | 39
    Hispanic or Latino Ethnicity | 18 | 23 | 41
NYHA Class [Count of Participants; unit: Participants] — Measure Description:
  New York Heart Association (NYHA) Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
  Participants
    I | 0 | 0 | 0
    II | 344 | 333 | 677
    III | 472 | 411 | 883
    IV | 48 | 52 | 100
Body Surface Area [Mean (Standard Deviation); unit: meters squared] — Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
  meters squared | 1.9 (0.2) | 1.9 (0.2) | 1.9 (0.2)
STS Score [Mean (Standard Deviation); unit: % risk of mortality] — Measure Description: The Society of Thoracic Surgeons (STS) risk model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. After information has been entered on a given case, the online STS risk calculator provides a risk percentage for each of the outcomes. The risk percentage estimates the chance of a specific outcome for a patient with the indicated risk factors. A higher score indicates a higher risk. A lower score indicates a lower risk.
  % risk of mortality | 4.4 (1.5) | 4.5 (1.6) | 4.5 (1.6)
Logistic EuroSCORE [Mean (Standard Deviation); unit: percentage of predicted mortality] — Measure Description: The European System for Cardiac Operative Risk Evaluation (EuroSCORE) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. A higher score indicates a higher risk. A lower score indicates a lower risk. Population: Data missing for 1 SAVR subject.
  percentage of predicted mortality
    number analyzed (Participants) | 864 | 795 | 1659
    (all) | 11.9 (7.6) | 11.6 (8.0) | 11.8 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality or Disabling Stroke Rate Expressed as a Posterior Probability
Description: All-cause mortality: all deaths from any cause after valve intervention. This includes all cardiovascular and non-cardiovascular deaths.
  Disabling Stroke: a modified rankin (mRS) score of 2 or more at 90 days and an increase in at least one mRS category from an individual's pre-strike baseline.
Time Frame: 24 months
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Median (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
Percentage of Participants | 12.6 [10.2 to 15.3] | 14.0 [11.4 to 17.0]
Statistical Analysis 1: Comparison: Medtronic CoreValve® System TAVI vs SAVR; Primary Hypothesis: TAVR with the Medtronic TAVR is non-inferior to SAVR for all-cause mortality or disabling stroke rate during a fixed follow-up of 24 months; Test type: Non-Inferiority — Non-inferiority margin was 0.07. Posterior threshold for non-inferiority was 0.971; Bayesian — The posterior probability of non-inferiority is > 0.9999. The posterior probability is the probability of the event rate by updating the prior probability distribution with observed data using Bayes' Theorem; Posterior Median of the Difference = -1.4 — 95% Bayesian credible interval for the difference (TAVR-SAVR) was (-5.2%, 2.3%). The 95% credible interval is the 2.5th and 97.5th percentiles of the posterior distribution

2. Secondary Outcome: Percentage of Participants With Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)
Description: MACCE is defined as a composite of:
  * All-cause death
  * Myocardial infarction (MI)
  * All stroke, and
  * Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 days | 5.7 | 7.3
  6 months | 9.5 | 10.7
  12 months | 13.0 | 13.0
  18 months | 15.6 | 14.8
  24 months | 18.5 | 18.2

3. Secondary Outcome: Percentage of Participants With Individual MACCE Components
Description: as for outcome 2
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 day All Cause Mortality | 2.1 | 1.6
  30 day MI | 0.8 | 0.9
  30 day Stroke | 3.3 | 5.4
  30 day Reintervention | 0.8 | 0.1
  6 month All Cause Mortality | 4.2 | 4.7
  6 month MI | 1.2 | 1.4
  6 month Stroke | 4.6 | 6.6
  6 month Reintervention | 1.8 | 0.3
  12 month All Cause Mortality | 6.5 | 6.7
  12 month MI | 1.9 | 1.4
  12 month Stroke | 5.2 | 6.9
  12 month Reintervention | 2.0 | 0.5
  18 month All Cause Mortality | 8.5 | 7.9
  18 month MI | 2.2 | 1.8
  18 month Stroke | 5.7 | 7.5
  18 month Reintervention | 2.4 | 0.5
  24 month All Cause Mortality | 11.5 | 10.5
  24 month MI | 2.7 | 2.2
  24 month Stroke | 6.0 | 8.5
  24 month Reintervention | 2.4 | 0.5

4. Secondary Outcome: Percentage of Participants With Major Adverse Events (MAE)
Description: Major Adverse Events (MAE) include all death, MI, all stroke, reintervention, cardiac perforation, cardiac tamponade, cardiogenic shock, valve malpositioning, prosthetic valve dysfunction, acute kidney injury, major vascular complication, life threatening or disabling bleed, major bleed, and valve endocarditis.
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 days | 23.7 | 30.3
  6 months | 28.5 | 33.6
  12 months | 33.0 | 35.8
  18 months | 36.6 | 38.4
  24 months | 40.0 | 41.8

5. Secondary Outcome: Percentage of Participants With Conduction Disturbance Requiring Permanent Pacemaker Implantation
Time Frame: 30 day, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 days | 25.6 | 6.5
  6 months | 27.2 | 7.6
  12 months | 28.3 | 8.6
  18 months | 30.1 | 9.2
  24 months | 30.9 | 9.8

6. Secondary Outcome: Change in NYHA Class From Baseline
Description: Change from baseline (continuous variable). A positive number corresponds to NYHA worsening; a negative number corresponds to NYHA improvement.
  New York Heart Association (NYHA) Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: Baseline to 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
units on a scale
  30 day | -1.2 (0.8) | -1.0 (0.9)
  6 month | -1.3 (0.8) | -1.3 (0.8)
  12 month | -1.3 (0.8) | -1.3 (0.8)
  18 month | -1.2 (0.8) | -1.2 (0.8)
  24 month | -1.2 (0.8) | -1.2 (0.8)

7. Secondary Outcome: Change in Distance Walked During 6-minute Walk Test (6MWT)
Description: Change in distance walked during 6MWT from baseline
Time Frame: From baseline to 30 days, baseline to 12 months, and baseline to 24 months
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
meters
  30 days | 35.4 (99.2) | -14.4 (108.7)
  12 months | 37.1 (103.5) | 17.8 (102.0)
  24 months | 26.5 (115.4) | 11.7 (102.7)

8. Secondary Outcome: Ratio of Days Alive Out of Hospital Versus Total Days Alive
Time Frame: 12 and 24 months
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
ratio
  12 months | 0.96 (0.12) | 0.93 (0.15)
  24 months | 0.96 (0.12) | 0.95 (0.15)

9. Secondary Outcome: Quality of Life (QoL) Change From Baseline
Description: QoL summary score change from baseline using the following measures:
  * Kansas City Cardiomyopathy Questionnaire (KCCQ): Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * 36 Item Short Form Health Survey (SF-36): Measures functional health and well-being. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * European QoL (EQ-5D): Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state.
Time Frame: Baseline, 30 days, 3 months, 6 months, 12 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
units on a scale
  30 day KCCQ- Overall | 18.4 (22.8) | 5.9 (27.0)
  30 day KCCQ- Clinical | 14.9 (21.2) | 4.0 (26.0)
  30 day SF-36-Physical | 5.7 (10.4) | -1.1 (11.0)
  30 day SF-36-Mental | 2.6 (12.3) | -0.6 (13.7)
  30 day EQ-5D | 0.06 (0.18) | -0.02 (0.21)
  3 month SF-36-Physical | 7.4 (10.5) | 5.6 (10.5)
  3 month SF-36-Mental | 4.6 (11.7) | 4.6 (12.6)
  3 month EQ-5D | 0.06 (0.18) | 0.05 (0.18)
  6 month KCCQ- Overall | 21.9 (22.3) | 21.3 (22.3)
  6 month KCCQ- Clinical | 16.5 (21.5) | 15.9 (21.7)
  6 month SF-36-Physical | 6.3 (10.3) | 6.3 (10.5)
  6 month SF-36-Mental | 3.9 (11.4) | 3.6 (11.9)
  6 month EQ-5D | 0.04 (0.18) | 0.05 (0.17)
  12 month KCCQ- Overall | 20.6 (22.3) | 20.5 (22.2)
  12 month KCCQ- Clinical | 15.1 (21.4) | 14.8 (21.6)
  12 month SF-36-Physical | 5.2 (9.9) | 5.2 (10.2)
  12 month SF-36-Mental | 4.0 (11.3) | 4.1 (12.0)
  12 month EQ-5D | 0.04 (0.16) | 0.03 (0.18)
  18 month KCCQ- Overall | 19.7 (21.5) | 20.2 (22.1)
  18 month KCCQ- Clinical | 14.0 (20.7) | 14.0 (21.9)
  18 month SF-36-Physical | 4.2 (10.4) | 4.3 (10.8)
  18 month SF-36-Mental | 4.3 (11.1) | 3.8 (11.9)
  18 month EQ-5D | 0.03 (0.17) | 0.03 (0.17)
  24 month KCCQ- Overall | 18.9 (21.2) | 18.6 (22.9)
  24 month KCCQ- Clinical | 12.7 (20.5) | 12.3 (22.5)
  24 month SF-36-Physical | 3.9 (9.9) | 4.0 (10.8)
  24 month SF-36-Mental | 3.6 (11.3) | 3.7 (12.2)
  24 month EQ-5D | 0.02 (0.17) | 0.02 (0.19)

10. Secondary Outcome: Transvalvular Mean Gradient (in mmHg) as an Assessment of Prosthetic Valve Performance
Description: Using the following measure:
  -Transvalvular mean gradient
Time Frame: discharge, 6 months, 12 months, and 24 months. Data for 3-5 years will be posted once data is complete
Population: Participant Population= Consisted of all randomized subjects with a valve implanted
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 863 | 794
mmHg
  discharge | 8.82 (3.89) | 12.39 (5.71)
  6 months | 8.28 (3.88) | 11.10 (4.72)
  12 months | 8.34 (3.89) | 11.57 (5.16)
  24 months | 8.20 (3.85) | 11.55 (5.43)

11. Secondary Outcome: Effective Orifice Area as an Assessment of Prosthetic Valve Performance
Description: Using the following measure:
  -Effective Orifice Area (cm^2)
Time Frame: discharge, 6 months, 12 months, and 24 months. Data for 3-5 years will be posted once data is complete
Population: Participant Population= Consisted of all randomized subjects with a valve implanted
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 863 | 794
cm^2
  discharge EOA | 2.13 (0.57) | 1.82 (0.63)
  6 months EOA | 2.14 (0.61) | 1.80 (0.57)
  12 months EOA | 2.13 (0.59) | 1.78 (0.59)
  24 months EOA | 2.15 (0.63) | 1.77 (0.55)

12. Secondary Outcome: Degree of Aortic Valve Regurgitation as an Assessment of Prosthetic Valve Performance
Description: Using the following measure:
  - Degree of Aortic Valve Regurgitation (Transvalvular and Paravalvular)
Time Frame: discharge, 6 months, 12 months, and 24 months. Data for 3-5 years will be posted once data is complete
Population: Participant Population= Consisted of all randomized subjects with a valve implanted
Measure: Number; unit: Percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 863 | 794
Percentage of participants
  Discharge : Total Aortic Regurgitation- None | 24.9 | 67.9
  Discharge : Total Aortic Regurgitation- Trace | 35.7 | 24.6
  Discharge : Total Aortic Regurgitation- Mild | 35.9 | 6.8
  Discharge : Total Aortic Regurgitation- Moderate | 3.2 | 0.7
  Discharge : Total Aortic Regurgitation- Severe | 0.2 | 0.0
  6 months : Total Aortic Regurgitation- None | 28.4 | 67.0
  6 months : Total Aortic Regurgitation- Trace | 32.2 | 24.3
  6 months : Total Aortic Regurgitation- Mild | 34.7 | 7.8
  6 months : Total Aortic Regurgitation- Moderate | 4.6 | 0.8
  6 months : Total Aortic Regurgitation- Severe | 0.1 | 0.2
  12 months : Total Aortic Regurgitation- None | 32.0 | 67.6
  12 months : Total Aortic Regurgitation- Trace | 28.8 | 23.5
  12 months : Total Aortic Regurgitation- Mild | 34.1 | 8.3
  12 months : Total Aortic Regurgitation- Moderate | 5.1 | 0.7
  12 months : Total Aortic Regurgitation- Severe | 0.0 | 0.0
  24 months : Total Aortic Regurgitation- None | 35.1 | 67.7
  24 months : Total Aortic Regurgitation- Trace | 30.5 | 25.3
  24 months : Total Aortic Regurgitation- Mild | 30.0 | 6.2
  24 months : Total Aortic Regurgitation- Moderate | 4.2 | 0.6
  24 months : Total Aortic Regurgitation- Severe | 0.2 | 0.2

13. Secondary Outcome: Percentage of Participants With Aortic Valve Disease Related Hospitalizations
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of particpants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of particpants
  30 days | 2.8 | 4.1
  6 months | 6.6 | 5.8
  12 months | 8.6 | 7.4
  18 months | 10.8 | 8.4
  24 months | 12.8 | 9.5

14. Secondary Outcome: Percentage of Participants With Cardiovascular Deaths and Valve-Related Deaths
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 day cardiovascular deaths | 2.0 | 1.6
  30 day valve related deaths | 0.0 | 0.0
  6 month cardiovascular deaths | 3.2 | 3.9
  6 month valve related deaths | 0.0 | 0.1
  12 month cardiovascular deaths | 4.7 | 5.3
  12 month valve related deaths | 0.0 | 0.1
  18 month cardiovascular deaths | 5.9 | 6.1
  18 month valve related deaths | 0.0 | 0.1
  24 month cardiovascular deaths | 7.8 | 7.1
  24 month valve related deaths | 0.0 | 0.1

15. Secondary Outcome: Percentage of Participants With Stroke and TIAs
Description: Strokes (of any severity) and Transient Ischemic Attacks (TIAs)
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 days | 4.4 | 6.3
  6 months | 6.9 | 7.8
  12 months | 8.0 | 8.6
  18 months | 8.8 | 9.4
  24 months | 9.5 | 11.2

16. Secondary Outcome: Peri-procedural Neurological Injury
Description: Neurological injury (stroke, TIA, or encephalopathy)
Time Frame: discharge or 7 days post index procedure (whichever occurred first)
Population: Participant Population= Consisted of all randomized subjects with an index procedure
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 863 | 795
percentage of participants | 4.8 | 12.3

17. Secondary Outcome: Index Procedure Related Major Adverse Events (MAEs)
Description: Index procedure related MAEs were defined as events occurring during, or as a direct result of, the index procedure.
Time Frame: Procedure through 30 day visit
Population: Participant Population= Consisted of all randomized subjects with an index procedure
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 863 | 795
percentage of participants | 23.5 | 30.4

18. Secondary Outcome: Length of Index Procedure Hospital Stay
Time Frame: Number of days from admission to discharge (expected average of 7 days)
Population: Participant Population= Consisted of all randomized subjects with an index procedure
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 863 | 795
days | 5.7 (4.9) | 9.8 (8.0)

19. Secondary Outcome: Presence of Atrial Fibrillation
Time Frame: post-procedure, discharge, 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  post procedure | 12.8 | 8.7
  discharge | 14.0 | 22.2
  30 days | 13.6 | 14.4
  6 months | 14.1 | 12.1
  12 months | 13.4 | 11.7
  18 months | 13.6 | 11.9
  24 months | 15.1 | 12.2

20. Secondary Outcome: Device Success (Medtronic CoreValve® System Subjects Only)
Description: * Absence of procedural mortality
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation)
Time Frame: Number of days from admission to discharge (expected average of 7 days)
Population: Participant Population =Consisted of all randomized subjects with a TAVR index procedure who were evaluable for device success.
Measure: Number; unit: percentage of participants
Groups:
- Medtronic CoreValve® System TAVI: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Medtronic CoreValve® Evolut R System Transcatheter Aortic Valve Implantation (TAVI)
Arm/Group | Medtronic CoreValve® System TAVI
Number analyzed (Participants) | 863
percentage of participants | 77.0

21. Secondary Outcome: Procedural Success (Medtronic CoreValve® System Subjects Only)
Description: Defined by device success and absence of in-hospital major adverse cardiovascular and cerebrovascular events (MACCE)
Time Frame: Number of days from admission to discharge (expected average of 7 days)
Population: Participant Population= Consisted of all randomized subjects with a TAVR index procedure who were evaluable for procedural success.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI
Number analyzed (Participants) | 863
percentage of participants | 74.7

22. Secondary Outcome: Evidence of Prosthetic Valve Dysfunction (Medtronic CoreValve® System Subjects Only)
Description: Prosthetic Valve Dysfunction (PVD) was defined according to Valve Academic Research Consortium (VARC) II using the Core Lab Echocardiography assessments including aortic regurgitation (AR) and aortic stenosis (AS) evaluations. Total aortic regurgitation (AR) reported as moderate or severe was considered
  PVD defined as:
  * Mean aortic valve gradient ≥20 mmHg AND ((EOA ≤0.9 cm2 if BSA <1.6 or ≤1.1 cm2 if BSA ≥1.6) OR DVI <0. 35 m/s) OR
  * moderate or severe total AR
Time Frame: 6 months, 12 months, and 24 months. Data for 3-5 years will be posted once data is complete.
Population: Participant Population= Consisted of all subjects with a valve implanted
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  6 month | 6.0 | 4.1
  12 month | 6.7 | 6.4
  24 month | 6.0 | 5.8

23. Secondary Outcome: Percentage of Participants With Early Safety Endpoint
Description: Percentage of participants with VARC II early safety composite at 30 days
Time Frame: 30 Days
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants | 12.5 | 15.8

24. Secondary Outcome: Percentage of Participants With Clinical Efficacy (After 30 Days)
Description: Combined clinical efficacy after 30 days was defined as the composite of all-cause mortality, all strokes (disabling and non-disabling), hospitalization for valve-related symptoms or worsening congestive heart failure, NYHA III or IV, and valve-related dysfunction.
Time Frame: 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is complete
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  6 months | 12.8 | 9.9
  12 months | 23.5 | 21.0
  18 months | 26.3 | 22.6
  24 months | 33.9 | 33.0

25. Secondary Outcome: Percentage of Participants With Time-Related Safety
Description: The VARC II time-related valve safety composite was defined as the rate of valve-related dysfunction (mean aortic valve gradient ≥ 20 mm Hg, EOA ≤ 0.9-1.1 cm2 depending on body surface area and/or DVI <0.35, AND/ OR moderate or severe prosthetic valve regurgitation), aortic valve reintervention, prosthetic valve endocarditis, prosthetic valve thrombosis, thromboembolic events, and VARC II bleeding events.
Time Frame: 30 days, 6 months, 12 months, 18 months, and 24 months. Data for 3-5 years will be posted once data is available.
Population: Participant Population= Consisted of all randomized subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
Number analyzed (Participants) | 864 | 796
percentage of participants
  30 days | 28.8 | 61.7
  6 months | 38.5 | 69.6
  12 months | 45.1 | 72.1
  18 months | 42.1 | 67.8
  24 months | 53.0 | 77.3

26. Secondary Outcome: Resheath and Recapture Success (Evolut R Only)
Description: The Evolut™ R system provides operators with the ability to resheath or recapture the valve before it is completely deployed in the event of initial suboptimal positioning. Successful resheath was defined as successfully retrieving a portion of the valve into the capsule of the delivery catheter, and successful recapture was defined as successfully recapturing the entirety of the valve into the capsule of the delivery catheter.
Time Frame: Procedure
Population: Participant Population= Consisted of all subjects in whom the resheath or recapture feature of the Evolut R system was attempted
Measure: Number; unit: percentage of attempts
Units Other Than Participants: attempts
Groups:
- Medtronic CoreValve® System TAVI: Medtronic CoreValve® Evolut R System Transcatheter Aortic Valve Implantation (TAVI)
Arm/Group | Medtronic CoreValve® System TAVI
Number analyzed (Participants) | 31
Number analyzed (attempts) | 53
percentage of attempts
  Resheath | 100
  Recapture | 89.7
  Resheath or Recapture | 92.5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study enrollment through the 24 month follow-up visit. Adverse event data are currently available and reported for up to 24 months.
Description: All new or worsening AEs were collected through 24 months.
Arm/Group | Medtronic CoreValve® System TAVI | SAVR
All-Cause Mortality (participants affected / at risk) | 98/864 | 80/796
Serious Adverse Events (participants affected / at risk) | 718/864 | 694/796
Other Adverse Events (participants affected / at risk) | 803/864 | 754/796
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic CoreValve® System TAVI (N=864) | SAVR (N=796)
ANAEMIA (Blood and lymphatic system disorders) | 102 (117) | 203 (222)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
BLOOD DISORDER (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
COAGULOPATHY (Blood and lymphatic system disorders) | 6 (6) | 11 (11)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 40 (40) | 84 (87)
HYPOCHROMIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 4 (4) | 7 (8)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
SPLENIC HAEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 10 (10) | 44 (45)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 0 (0)
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 12 (12) | 9 (15)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 17 (17) | 19 (19)
ANGINA PECTORIS (Cardiac disorders) | 11 (11) | 4 (5)
ANGINA UNSTABLE (Cardiac disorders) | 4 (4) | 3 (3)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1) | 1 (1)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 43 (46) | 5 (5)
AORTIC VALVE STENOSIS (Cardiac disorders) | 2 (2) | 4 (5)
ARRHYTHMIA (Cardiac disorders) | 3 (3) | 3 (3)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 86 (105) | 169 (185)
ATRIAL FLUTTER (Cardiac disorders) | 10 (11) | 19 (19)
ATRIAL RUPTURE (Cardiac disorders) | 0 (0) | 2 (2)
ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 4 (4)
ATRIAL THROMBOSIS (Cardiac disorders) | 2 (2) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 18 (18) | 5 (5)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 157 (157) | 44 (44)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 16 (16) | 2 (2)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 17 (18) | 6 (6)
ATRIOVENTRICULAR DISSOCIATION (Cardiac disorders) | 2 (2) | 0 (0)
BRADYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 27 (27) | 17 (18)
BUNDLE BRANCH BLOCK (Cardiac disorders) | 1 (1) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 58 (58) | 1 (1)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 7 (8) | 3 (3)
CARDIAC ARREST (Cardiac disorders) | 21 (21) | 15 (15)
CARDIAC FAILURE (Cardiac disorders) | 21 (28) | 21 (27)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 10 (11) | 6 (6)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 3 (3) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 82 (104) | 61 (74)
CARDIAC PERFORATION (Cardiac disorders) | 12 (13) | 1 (1)
CARDIAC SEPTAL HYPERTROPHY (Cardiac disorders) | 1 (1) | 2 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 12 (12) | 9 (9)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 6 (6) | 5 (5)
CARDIOGENIC SHOCK (Cardiac disorders) | 9 (9) | 32 (32)
CARDIOMYOPATHY (Cardiac disorders) | 2 (2) | 3 (3)
CARDIORENAL SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOVASCULAR DECONDITIONING (Cardiac disorders) | 0 (0) | 3 (3)
CHRONOTROPIC INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
CONDUCTION DISORDER (Cardiac disorders) | 3 (3) | 0 (0)
COR PULMONALE (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 6 (6) | 5 (5)
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 2 (2) | 1 (1)
CORONARY OSTIAL STENOSIS (Cardiac disorders) | 1 (1) | 1 (1)
DEFECT CONDUCTION INTRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1)
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
DRESSLER'S SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 1 (1)
INTRAPERICARDIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 0 (0)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 3 (3)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 2 (2) | 5 (5)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 3 (3) | 4 (4)
LOW CARDIAC OUTPUT SYNDROME (Cardiac disorders) | 0 (0) | 4 (4)
MITRAL VALVE CALCIFICATION (Cardiac disorders) | 0 (0) | 1 (1)
MITRAL VALVE DISEASE MIXED (Cardiac disorders) | 0 (0) | 1 (1)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 10 (11) | 6 (6)
MITRAL VALVE STENOSIS (Cardiac disorders) | 0 (0) | 3 (3)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4) | 4 (4)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 3 (3)
NODAL ARRHYTHMIA (Cardiac disorders) | 3 (3) | 1 (1)
NODAL RHYTHM (Cardiac disorders) | 5 (5) | 6 (6)
PALPITATIONS (Cardiac disorders) | 0 (0) | 3 (3)
PARAVALVULAR AORTIC REGURGITATION (Cardiac disorders) | 7 (7) | 0 (0)
PAROXYSMAL ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 12 (12) | 15 (16)
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 (1) | 2 (2)
PERICARDITIS (Cardiac disorders) | 0 (0) | 5 (5)
PROSTHETIC CARDIAC VALVE THROMBOSIS (Cardiac disorders) | 1 (1) | 3 (3)
PULMONARY VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 1 (1)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 2 (2) | 3 (3)
RHYTHM IDIOVENTRICULAR (Cardiac disorders) | 1 (1) | 1 (1)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 2 (2)
RIGHT VENTRICULAR ENLARGEMENT (Cardiac disorders) | 0 (0) | 1 (1)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 4 (4) | 4 (4)
SINUS ARREST (Cardiac disorders) | 2 (2) | 2 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 3 (3)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 9 (9) | 9 (10)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2) | 3 (3)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 7 (7) | 5 (5)
SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 6 (6) | 3 (3)
TORSADE DE POINTES (Cardiac disorders) | 0 (0) | 1 (1)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 8 (8) | 12 (12)
TRIFASCICULAR BLOCK (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR ASYSTOLE (Cardiac disorders) | 1 (1) | 1 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 3 (3) | 3 (3)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 5 (5) | 7 (7)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 15 (17) | 15 (16)
HAEMOPHILIA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
LEFT VENTRICLE OUTFLOW TRACT OBSTRUCTION (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
CERUMEN IMPACTION (Ear and labyrinth disorders) | 1 (1) | 1 (1)
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 3 (3) | 2 (2)
GOITRE (Endocrine disorders) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM PRIMARY (Endocrine disorders) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 2 (2)
AMAUROSIS FUGAX (Eye disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 10 (11) | 7 (9)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 1 (1)
CHARLES BONNET SYNDROME (Eye disorders) | 1 (1) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
DIABETIC RETINAL OEDEMA (Eye disorders) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
MACULAR FIBROSIS (Eye disorders) | 0 (0) | 1 (1)
OPEN ANGLE GLAUCOMA (Eye disorders) | 0 (0) | 1 (1)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 1 (1)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 4 (4)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 3 (3)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 2 (2) | 1 (1)
ANAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 2 (3) | 0 (0)
COLITIS (Gastrointestinal disorders) | 3 (3) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 2 (2) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 3 (4)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 7 (7)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 4 (4)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DYSKINESIA OESOPHAGEAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 10 (10) | 22 (22)
FAECALOMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 24 (28) | 28 (34)
GASTROINTESTINAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 3 (3)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
ILEUS (Gastrointestinal disorders) | 4 (4) | 4 (4)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 2 (2)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INCARCERATED UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 4 (4) | 3 (3)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 2 (3) | 2 (2)
INTESTINAL MASS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1) | 2 (2)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 3 (4) | 1 (1)
LOOSE TOOTH (Gastrointestinal disorders) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 6 (7) | 3 (3)
MELAENA (Gastrointestinal disorders) | 1 (1) | 4 (4)
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2)
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERITONEAL LESION (Gastrointestinal disorders) | 1 (1) | 0 (0)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 4 (4) | 4 (4)
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTOURETHRAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 2 (2) | 1 (1)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
SALIVARY GLAND MASS (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 3 (3)
SWOLLEN TONGUE (Gastrointestinal disorders) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 3 (3)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 4 (4)
VOLVULUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (3) | 4 (4)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 2 (2)
ASTHENIA (General disorders) | 9 (9) | 7 (9)
CATHETER SITE DISCHARGE (General disorders) | 1 (1) | 2 (2)
CATHETER SITE HAEMATOMA (General disorders) | 1 (1) | 0 (0)
CATHETER SITE HAEMORRHAGE (General disorders) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 2 (2) | 2 (2)
CHEST PAIN (General disorders) | 18 (20) | 17 (18)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 1 (1) | 1 (1)
COMPLICATION OF DEVICE INSERTION (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 5 (5) | 4 (4)
DEVICE EMBOLISATION (General disorders) | 2 (2) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 1 (1)
EFFUSION (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1)
GAIT DISTURBANCE (General disorders) | 4 (4) | 1 (1)
GENERALISED OEDEMA (General disorders) | 0 (0) | 1 (1)
HERNIA (General disorders) | 0 (0) | 1 (1)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 1 (1)
IMPLANT SITE DISCHARGE (General disorders) | 0 (0) | 1 (1)
IMPLANT SITE EROSION (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 2 (2) | 5 (5)
NON-CARDIAC CHEST PAIN (General disorders) | 7 (7) | 12 (13)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 11 (12)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1)
POLYP (General disorders) | 2 (2) | 0 (0)
PUNCTURE SITE HAEMORRHAGE (General disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 8 (8)
SUDDEN CARDIAC DEATH (General disorders) | 2 (2) | 0 (0)
SUDDEN DEATH (General disorders) | 1 (1) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 (2) | 6 (6)
ULCER HAEMORRHAGE (General disorders) | 0 (0) | 1 (1)
VASCULAR STENT STENOSIS (General disorders) | 0 (0) | 1 (1)
VASCULAR STENT THROMBOSIS (General disorders) | 1 (1) | 0 (0)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 3 (3) | 1 (1)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2) | 4 (4)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 2 (2)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2) | 5 (5)
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
GALLBLADDER DISORDER (Hepatobiliary disorders) | 0 (0) | 2 (2)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 (1) | 2 (2)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (2) | 0 (0)
ABSCESS JAW (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
ARTHRITIS INFECTIVE (Infections and infestations) | 1 (1) | 1 (1)
BACTERAEMIA (Infections and infestations) | 12 (13) | 4 (4)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 6 (6) | 5 (5)
CAMPYLOBACTER SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
CARDIAC VALVE ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
CATHETER SITE CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 16 (17) | 15 (15)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 3 (3) | 5 (5)
CYSTITIS (Infections and infestations) | 0 (0) | 2 (2)
CYTOMEGALOVIRUS VIRAEMIA (Infections and infestations) | 1 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (1) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 4 (4) | 0 (0)
EMPYEMA (Infections and infestations) | 1 (1) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 1 (1)
ENCEPHALITIS VIRAL (Infections and infestations) | 0 (0) | 2 (2)
ENDOCARDITIS (Infections and infestations) | 6 (6) | 8 (8)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ENTEROBACTER SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 3 (4) | 0 (0)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
EPIDIDYMITIS (Infections and infestations) | 1 (1) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 2 (2) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
FUNGAL OESOPHAGITIS (Infections and infestations) | 1 (1) | 0 (0)
GANGRENE (Infections and infestations) | 0 (0) | 3 (3)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
GROIN INFECTION (Infections and infestations) | 2 (2) | 1 (1)
HAEMOPHILUS SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
HELICOBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 2 (2)
INCISION SITE CELLULITIS (Infections and infestations) | 1 (1) | 1 (1)
INFECTED SEROMA (Infections and infestations) | 0 (0) | 1 (2)
INFECTION (Infections and infestations) | 2 (2) | 3 (3)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 1 (1)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 2 (2) | 1 (1)
LABYRINTHITIS (Infections and infestations) | 0 (0) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0)
LIVER ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 2 (2) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (2)
LYME DISEASE (Infections and infestations) | 0 (0) | 1 (1)
MEDIASTINITIS (Infections and infestations) | 1 (1) | 2 (2)
NASAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ORCHITIS (Infections and infestations) | 2 (2) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 3 (3) | 4 (7)
OSTEOMYELITIS ACUTE (Infections and infestations) | 0 (0) | 2 (3)
PERITONITIS (Infections and infestations) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 58 (65) | 55 (60)
PNEUMONIA BACTERIAL (Infections and infestations) | 4 (5) | 2 (2)
PNEUMONIA CYTOMEGALOVIRAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 1 (1)
POST PROCEDURAL PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 6 (6) | 13 (19)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
PSEUDOMONAS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 1 (1) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 1 (1)
RESPIRATORY SYNCYTIAL VIRUS BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 5 (5)
SALMONELLA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 24 (28) | 24 (25)
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 0 (0) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 5 (5) | 5 (6)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1)
SKIN CANDIDA (Infections and infestations) | 0 (0) | 1 (1)
SPINAL CORD INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 2 (2)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 2 (3) | 0 (0)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 33 (41) | 25 (26)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 8 (10) | 12 (12)
VASCULAR ACCESS SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VIRAL CARDIOMYOPATHY (Infections and infestations) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 2 (2)
WOUND INFECTION (Infections and infestations) | 1 (1) | 4 (4)
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 17 (17) | 36 (36)
ANASTOMOTIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
AORTIC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTERIAL BYPASS OCCLUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
BRACHIAL PLEXUS INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC VALVE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CARDIAC VEIN PERFORATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COMPLICATIONS OF TRANSPLANTED HEART (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
DEVICE DEPLOYMENT ISSUE (Injury, poisoning and procedural complications) | 24 (25) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 13 (14) | 9 (9)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOREIGN BODY IN EAR (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAEMODILUTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
HEART INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 11 (11) | 10 (10)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
INCISIONAL HERNIA, OBSTRUCTIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
JOINT INJURY (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
LACERATION (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PERIPROCEDURAL MYOCARDIAL INFARCTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 19 (20)
POSTOPERATIVE DELIRIUM (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
POSTOPERATIVE RESPIRATORY FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
POSTOPERATIVE THORACIC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
POSTOPERATIVE THROMBOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (2) | 9 (9)
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
PROCEDURAL PNEUMOTHORAX (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN ABRASION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC LUNG INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
URETERIC INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
URINARY RETENTION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VASCULAR ACCESS SITE COMPLICATION (Injury, poisoning and procedural complications) | 9 (9) | 0 (0)
VASCULAR ACCESS SITE HAEMATOMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
VASCULAR ACCESS SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 7 (7) | 2 (2)
VASOPLEGIA SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VENOUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WEANING FAILURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
WOUND SECRETION (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
XIITH NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANTICOAGULATION DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 2 (2) | 5 (5)
ANTICOAGULATION DRUG LEVEL BELOW THERAPEUTIC (Investigations) | 0 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 3 (3) | 0 (0)
BLOOD CULTURE POSITIVE (Investigations) | 1 (1) | 1 (1)
BLOOD ERYTHROPOIETIN DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD FIBRINOGEN DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD POTASSIUM ABNORMAL (Investigations) | 1 (1) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 1 (1) | 0 (0)
BRAIN NATRIURETIC PEPTIDE INCREASED (Investigations) | 0 (0) | 2 (2)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1)
CALCIUM IONISED DECREASED (Investigations) | 1 (1) | 0 (0)
CARDIAC INDEX DECREASED (Investigations) | 1 (1) | 3 (3)
CARDIAC INDEX INCREASED (Investigations) | 0 (0) | 1 (1)
CARDIAC MURMUR (Investigations) | 0 (0) | 1 (1)
CARDIAC OUTPUT DECREASED (Investigations) | 1 (1) | 9 (9)
CARDIOVASCULAR FUNCTION TEST NORMAL (Investigations) | 0 (0) | 1 (1)
COAGULATION TIME PROLONGED (Investigations) | 0 (0) | 2 (2)
CYSTOSCOPY ABNORMAL (Investigations) | 1 (1) | 0 (0)
ECHOCARDIOGRAM ABNORMAL (Investigations) | 0 (0) | 3 (3)
EJECTION FRACTION DECREASED (Investigations) | 3 (3) | 1 (1)
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 2 (2) | 0 (0)
ELECTROCARDIOGRAM ST SEGMENT ABNORMAL (Investigations) | 0 (0) | 1 (1)
FIBRIN D DIMER INCREASED (Investigations) | 0 (0) | 1 (1)
FUNGAL TEST POSITIVE (Investigations) | 0 (0) | 1 (1)
HAEMATOCRIT DECREASED (Investigations) | 0 (0) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 6 (6) | 5 (5)
INTERNATIONAL NORMALISED RATIO ABNORMAL (Investigations) | 0 (0) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 5 (5)
INVESTIGATION (Investigations) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
NUTRITIONAL CONDITION ABNORMAL (Investigations) | 0 (0) | 1 (1)
OCCULT BLOOD (Investigations) | 0 (0) | 1 (1)
OCCULT BLOOD POSITIVE (Investigations) | 1 (1) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 2 (2)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
PULMONARY ARTERIAL PRESSURE ABNORMAL (Investigations) | 1 (1) | 0 (0)
PULSE ABSENT (Investigations) | 1 (1) | 0 (0)
TROPONIN INCREASED (Investigations) | 4 (4) | 1 (1)
URINE OUTPUT DECREASED (Investigations) | 5 (5) | 3 (3)
VENOUS OXYGEN SATURATION ABNORMAL (Investigations) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 2 (2)
WEIGHT INCREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1 (1) | 2 (2)
ABNORMAL LOSS OF WEIGHT (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
CALCIPHYLAXIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (8) | 5 (5)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 13 (14) | 29 (29)
GOUT (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 10 (10) | 14 (14)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 7 (7)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 (6) | 8 (9)
HYPOMAGNEseriousMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 12 (14) | 16 (18)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 17 (17)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALNUTRITION (Metabolism and nutrition disorders) | 2 (2) | 9 (9)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
BURSITIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FISTULA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
JAW CYST (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 16 (17) | 12 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPONDYLOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TEMPOROMANDIBULAR JOINT SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENOSYNOVITIS STENOSANS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 7 (7)
BASOSQUAMOUS CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6)
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BONE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
CHRONIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GALLBLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTROINTESTINAL STROMAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LENTIGO MALIGNA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LIPOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
MALIGNANT NEOPLASM OF SPERMATIC CORD (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0)
APHASIA (Nervous system disorders) | 2 (2) | 2 (2)
BRAIN INJURY (Nervous system disorders) | 0 (0) | 1 (1)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 6 (6) | 4 (4)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 3 (4) | 1 (1)
CEREBELLAR HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBELLAR INFARCTION (Nervous system disorders) | 3 (3) | 1 (1)
CEREBRAL ATROPHY (Nervous system disorders) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 3 (3) | 7 (7)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 24 (25) | 30 (31)
COGNITIVE DISORDER (Nervous system disorders) | 2 (2) | 0 (0)
COMA (Nervous system disorders) | 0 (0) | 1 (1)
DEMENTIA (Nervous system disorders) | 1 (1) | 1 (1)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 3 (3) | 0 (0)
DIZZINESS (Nervous system disorders) | 8 (9) | 3 (3)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 1 (1)
EMBOLIC CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
EMBOLIC STROKE (Nervous system disorders) | 1 (1) | 2 (2)
ENCEPHALOPATHY (Nervous system disorders) | 6 (6) | 6 (7)
EPILEPSY (Nervous system disorders) | 2 (2) | 1 (1)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 2 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 (1) | 5 (5)
HAEMORRHAGIC STROKE (Nervous system disorders) | 4 (4) | 4 (4)
HEADACHE (Nervous system disorders) | 3 (3) | 0 (0)
HEMIANOPIA (Nervous system disorders) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 2 (2)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
HYPERREFLEXIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 1 (1)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 1 (1)
IIIRD NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 4 (4) | 8 (8)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
LETHARGY (Nervous system disorders) | 1 (1) | 2 (2)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 5 (5) | 7 (7)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 1 (1)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 2 (2) | 1 (1)
PERONEAL NERVE PALSY (Nervous system disorders) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 2 (2) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 9 (12) | 4 (4)
SEIZURE (Nervous system disorders) | 2 (2) | 1 (1)
SEIZURE LIKE PHENOMENA (Nervous system disorders) | 0 (0) | 1 (1)
SENSORY DISTURBANCE (Nervous system disorders) | 1 (1) | 0 (0)
SEROTONIN SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 24 (24) | 19 (20)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 25 (25) | 10 (10)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 1 (1) | 0 (0)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 1 (1)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
DEVICE ADHESION ISSUE (Product Issues) | 0 (0) | 2 (2)
DEVICE CAPTURING ISSUE (Product Issues) | 1 (1) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 3 (3) | 1 (1)
DEVICE FAILURE (Product Issues) | 1 (1) | 0 (0)
DEVICE ISSUE (Product Issues) | 1 (1) | 1 (1)
DEVICE LEAD ISSUE (Product Issues) | 0 (0) | 2 (2)
DEVICE LEAKAGE (Product Issues) | 28 (30) | 2 (2)
DEVICE LOOSENING (Product Issues) | 1 (1) | 0 (0)
DEVICE MALFUNCTION (Product Issues) | 1 (1) | 2 (2)
DEVICE PACING ISSUE (Product Issues) | 1 (1) | 0 (0)
LEAD DISLODGEMENT (Product Issues) | 6 (6) | 2 (2)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (2)
AGITATION (Psychiatric disorders) | 3 (3) | 3 (3)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 5 (5)
DELIRIUM (Psychiatric disorders) | 5 (5) | 15 (16)
DELIRIUM TREMENS (Psychiatric disorders) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 (1) | 0 (0)
DISORIENTATION (Psychiatric disorders) | 1 (1) | 0 (0)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 0 (0) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 13 (13) | 8 (8)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 62 (75) | 82 (95)
ANURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
AZOTAEMIA (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 6 (6) | 4 (4)
DYSURIA (Renal and urinary disorders) | 2 (2) | 1 (1)
END STAGE RENAL DISEASE (Renal and urinary disorders) | 1 (2) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 22 (25) | 15 (18)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 (0) | 1 (1)
INCONTINENCE (Renal and urinary disorders) | 2 (2) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (3) | 2 (3)
OLIGURIA (Renal and urinary disorders) | 3 (3) | 2 (2)
POLYURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY OCCLUSION (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 7 (8) | 13 (13)
RENAL HAEMORRHAGE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL MASS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL TUBULAR DISORDER (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
STAG HORN CALCULUS (Renal and urinary disorders) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 29 (32) | 21 (21)
URINE FLOW DECREASED (Renal and urinary disorders) | 1 (1) | 0 (0)
ACQUIRED PHIMOSIS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2 (2) | 1 (1)
PENILE OEDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PENILE PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE POLYP (Reproductive system and breast disorders) | 1 (1) | 1 (1)
ACUTE LUNG INJURY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 16 (16)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (11)
CHOKING SENSATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 16 (21)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
DEPENDENCE ON RESPIRATOR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 11 (11)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 10 (10)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (8)
LARYNGEAL ATROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
MEDIASTINAL HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
MEDIASTINAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8)
MEDIASTINAL MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 38 (43) | 102 (123)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 18 (18)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 10 (10)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PULMONARY HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 11 (11)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 50 (56)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
DIABETIC ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PANNICULITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CARDIAC PACEMAKER BATTERY REPLACEMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
CARDIAC PACEMAKER REPLACEMENT (Surgical and medical procedures) | 1 (1) | 1 (1)
CATARACT OPERATION (Surgical and medical procedures) | 1 (1) | 4 (5)
CHOLECYSTECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
COLOSTOMY CLOSURE (Surgical and medical procedures) | 0 (0) | 1 (1)
EAR OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 4 (4) | 0 (0)
IMPLANTABLE DEFIBRILLATOR REPLACEMENT (Surgical and medical procedures) | 0 (0) | 1 (1)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 2 (2)
PREVENTIVE SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
ROTATOR CUFF REPAIR (Surgical and medical procedures) | 1 (1) | 0 (0)
SPINAL FUSION SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1)
TRANSFUSION (Surgical and medical procedures) | 0 (0) | 1 (1)
WOUND DRAINAGE (Surgical and medical procedures) | 0 (0) | 2 (2)
WOUND TREATMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 1 (1) | 1 (1)
AORTIC ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1)
AORTIC DISSECTION (Vascular disorders) | 5 (6) | 0 (0)
AORTIC RUPTURE (Vascular disorders) | 1 (1) | 3 (3)
AORTIC STENOSIS (Vascular disorders) | 0 (0) | 1 (1)
ARTERIAL RUPTURE (Vascular disorders) | 2 (2) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 0 (0) | 4 (4)
ARTERY DISSECTION (Vascular disorders) | 1 (1) | 0 (0)
BRACHIOCEPHALIC VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 11 (11) | 11 (11)
DRY GANGRENE (Vascular disorders) | 0 (0) | 1 (1)
FEMORAL ARTERY DISSECTION (Vascular disorders) | 8 (8) | 2 (2)
FEMORAL ARTERY EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
FEMORAL ARTERY PERFORATION (Vascular disorders) | 3 (3) | 0 (0)
HAEMATOMA (Vascular disorders) | 24 (24) | 5 (5)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 3 (3) | 3 (3)
HAEMORRHAGE (Vascular disorders) | 17 (17) | 20 (20)
HYPERTENSION (Vascular disorders) | 34 (35) | 29 (32)
HYPERTENSIVE CRISIS (Vascular disorders) | 2 (4) | 3 (3)
HYPOTENSION (Vascular disorders) | 51 (52) | 87 (89)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 4 (4) | 10 (10)
ILIAC ARTERY PERFORATION (Vascular disorders) | 1 (1) | 0 (0)
ILIAC ARTERY RUPTURE (Vascular disorders) | 1 (1) | 0 (0)
INTERMITTENT CLAUDICATION (Vascular disorders) | 2 (2) | 0 (0)
LABILE BLOOD PRESSURE (Vascular disorders) | 3 (3) | 0 (0)
LYMPHOCELE (Vascular disorders) | 1 (1) | 0 (0)
MALIGNANT HYPERTENSION (Vascular disorders) | 2 (2) | 0 (0)
NECROSIS ISCHAEMIC (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 4 (4) | 7 (7)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (3) | 2 (2)
PERIPHERAL ARTERY DISSECTION (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 6 (6) | 0 (0)
PERIPHERAL ARTERY STENOSIS (Vascular disorders) | 12 (12) | 3 (3)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 5 (5) | 2 (3)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 2 (3) | 2 (2)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 1 (2) | 1 (1)
SHOCK (Vascular disorders) | 1 (1) | 7 (7)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 2 (2)
SUBCLAVIAN ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS (Vascular disorders) | 0 (0) | 2 (2)
VARICOSE VEIN (Vascular disorders) | 0 (0) | 1 (1)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic CoreValve® System TAVI (N=864) | SAVR (N=796)
ANAEMIA (Blood and lymphatic system disorders) | 80 (84) | 99 (100)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 70 (71) | 146 (154)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 133 (140) | 188 (198)
ATRIAL FIBRILLATION (Cardiac disorders) | 112 (120) | 230 (239)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 80 (82) | 67 (68)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 258 (265) | 55 (59)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 53 (56)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 42 (43)
OEDEMA PERIPHERAL (General disorders) | 45 (48) | 47 (49)
URINARY TRACT INFECTION (Infections and infestations) | 65 (77) | 88 (102)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 (0) | 122 (127)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 53 (54) | 102 (102)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 41 (42)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 46 (49) | 53 (55)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 52 (56)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 44 (47)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 79 (91) | 125 (138)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 62 (64) | 151 (154)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 48 (50) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 70 (76) | 216 (223)
HAEMATOMA (Vascular disorders) | 47 (49) | 0 (0)
HYPERTENSION (Vascular disorders) | 123 (139) | 100 (107)
HYPOTENSION (Vascular disorders) | 47 (50) | 82 (83)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT01586910/Prot_SAP_000.pdf